CLINICAL TRIAL: NCT03282513
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of AG-120 (Ivosidenib) in Subjects With Mild or Moderate Hepatic Impairment or Normal Hepatic Function
Brief Title: A Study of AG-120 (Ivosidenib) in Subjects With Mild or Moderate Hepatic Impairment or Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG120-C-012
Record Dates: First submitted 2017-09-08; First posted 2017-09-14 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Hepatic Impairment
Keywords: AG-120; Healthy Volunteer; Clinical Pharmacology; Hepatic Impairment
MeSH Terms: interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1A: Mild Hepatic Impairment (Experimental): Drug: AG-120 (Ivosidenib)
  A single 500 mg oral dose of AG-120 (Ivosidenib) in subjects with mild hepatic impairment(Child-Pugh Score A.)
  Interventions: Drug: AG-120 (Ivosidenib)
- Cohort 1B: Healthy Volunteers (Active Comparator): Drug: AG-120 (Ivosidenib)
  A single 500 mg oral dose of AG-120 (Ivosidenib) in subjects with normal hepatic function.
  Interventions: Drug: AG-120 (Ivosidenib)
- Cohort 2A: Moderate Hepatic Impairment (Experimental): Drug: AG-120 (Ivosidenib)
  A single 500 mg oral dose of AG-120 (Ivosidenib) in subjects with moderate hepatic impairment (Child-Pugh Score B.)
  Interventions: Drug: AG-120 (Ivosidenib)
- Cohort 2B: Healthy Volunteers (Active Comparator): Drug: AG-120 (Ivosidenib)
  A single 500 mg oral dose of AG-120 (Ivosidenib) in subjects with normal hepatic function.
  Interventions: Drug: AG-120 (Ivosidenib)

INTERVENTIONS:
Drug: AG-120 (Ivosidenib) — Single 500 mg dose of AG-120 (Ivosidenib).

SUMMARY:
Study AG120-C-012 is a Phase 1, open-label, single-dose study designed to evaluate the PK, safety, and tolerability of a single 500 mg AG-120 (Ivosidenib) dose in subjects with mild or moderate hepatic impairment (HI) compared to subjects with normal hepatic function. The study will be conducted at 2 US centers.

ELIGIBILITY:
Key Inclusion Criteria:

All subjects:

* Body Mass Index BMI of 19 to 40 kg/m2 (inclusive).
* Willing and able to comply with all study restrictions and requirements.
* Non- smoker, or uses no more nicotine-containing product than the equivalent of smoking ≤10 cigarettes per day, as judged by the investigator.
* Female subjects must be non pregnant and non-lactating and either be post-menopausal, surgically sterile, practice total abstinence from sexual intercourse as the preferred lifestyle or agree to use an appropriate method of birth control consistently throughout the study, from screening until 90 days after study drug administration.
* Male subjects with a partner of child bearing potential must either be sterile, practice total abstinence from sexual intercourse as the preferred life style or agree to use an appropriate method of birth control consistently throughout the study, from screening until 90 days after study drug administration.

Subjects with hepatic impairment (Cohorts 1a, 2a)

* Diagnosis of chronic (≥3 months prior to Screening) or stable (no acute episodes of illness within 2 months prior to Screening due to deterioration in hepatic function) hepatic insufficiency, with a Child-Pugh classification score in the mild or moderate range.
* Hepatic insufficiency may be of any etiology associated with an unambiguous medical history (such as evidence of portal hypertension).
* Other than hepatic insufficiency with features of cirrhosis, subjects are in good health based on medical history, physical exam, ECG, clinical laboratory tests, and Investigator's assessment.

Healthy matched subjects (Cohorts 1b, 2b)

• Have normal hepatic function and considered by the Investigator to be in good health, based on medical and surgical history review, physical exam, ECG, clinical laboratory tests, and Investigator's assessment.

Key Exclusion Criteria:

All subjects:

* Significant acute, new-onset illness (eg, flu, gastroenteritis) within 2 weeks prior to dosing.
* Positive test for drugs of abuse and/or positive alcohol test at Screening or prior to dosing.
* Medical history of clinically significant ECG abnormalities or a family history of prolonged QT interval syndromes.
* History of immunocompromise, including positivity for HIV, or active viral hepatitis B or C.
* Use of over the counter (OTC) medications, herbal supplements, grapefruit juice, Seville oranges, or vitamins 14 days prior to dosing.
* A recent (within 6 months prior to dosing) history of acute or chronic bronchospastic disease, including asthma and chronic obstructive pulmonary disease.
* Current or history of hepatic carcinoma, hepatorenal syndrome, portacaval shunt surgery, or pleural effusion. Malignancy, including leukemia and lymphoma, within the last 5 years.
* Any surgical or medical condition that might significantly alter the absorption, distribution, or excretion of AG-120.
* Treatment with strong cytochrome P450 (CYP)3A4 inhibitors or inducers within 14 days prior to AG 120 dosing or during the study.

Subjects with hepatic impairment (Cohorts 1a, 2a)

* Clinical evidence of moderate to severe ascites.
* Significant history or clinical manifestation of any significant metabolic/endocrine, allergic, dermatologic, renal, hematologic, pulmonary, immune, cardiovascular, gastrointestinal, genitourinary, neurologic, or psychiatric disorder, as determined by the Investigator and/or Sponsor's medical monitor (MM) to be clinically significant (CS.)
* Any evidence of progressive liver disease (within the last 4 weeks prior to dosing)
* Severe or uncontrolled medical conditions within 4 weeks prior to AG-120 dosing, with the exception of illness related to HI.

Healthy Matched Subjects

* Clinical evidence of liver disease or liver injury
* History or presence of impaired renal function
* QTCF >450 (males) or >460 (females) or ECG findings deemed abnormal by the Investigator
* Use of any prescription medications within 30 days prior to dosing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Predose; 0.5hr, 1hr, 2hr, 3hr, 4hr, 6hr, 9hr, 12hr, 24hr, 48hr, 72hr, 120hr, 168hr, 240hr, 336hr, and 504hr post dose
  AG-120 Cmax, derived from plasma concentration-time curves
Area under plasma concentration-time curve (AUC) | Predose; 0.5hr, 1hr, 2hr, 3hr, 4hr, 6hr, 9hr, 12hr, 24hr, 48hr, 72hr, 120hr, 168hr, 240hr, 336hr, and 504hr post dose
  AG-120 AUC, derived from plasma concentration-time curves

SECONDARY OUTCOMES:
Adverse Events (AE) and treatment-related AE | From the time of study drug administration through the end of study (Day 29 or early termination)
Plasma Protein Binding | Time Frame: Pre-dose, Day 1 and Day 2
  Compare the plasma protein binding of AG-120 (Ivosidenib) in subjects with impaired HI with that in subjects with normal hepatic function.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - DaVita Clinical Research- Colorado, Lakewood, Colorado
  - DaVita Clinical Research- Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] Fan B, Dai D, Cohen M, Xu H, Yin F, Nagaraja R, Mobilia M, Almon C, Basile FG, Yang H. Effect of Mild and Moderate Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of a Single Dose of Oral Ivosidenib in Otherwise Healthy Participants. Clin Pharmacol Drug Dev. 2021 Jan;10(1):99-109. doi: 10.1002/cpdd.821. Epub 2020 Jul 9. PMID 32648303